CLINICAL TRIAL: NCT04430478
Title: VOLume Flow-guided Angioplasty of Dysfunctional Autologous Arteriovenous Fistula. The VOLA Pilot Study
Brief Title: Volume Flow-guided Angioplasty of Dysfunctional Dialysis Access
Acronym: VOLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Stavros Spiliopoulos, Assistant Professor in Interventional Radiology, Attikon Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 323
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Dialysis Access Malfunction
Keywords: Percutaneous transluminal angioplasty; Volume-flow measurment; Autologous arteriovenous fistula; Dialysis access

STUDY DESIGN:
Intervention Model Description: The study will include consecutive patients undergoing fluoroscopically-guided percutaneous balloon angioplasty due to dysfunctional AVF. Intraprocedural volume flow measurements will be obtained just prior to the procedure and after each balloon dilation. Volume flow measurements will be correlated with digital subtraction angiography quantitative vessel analysis (QVA) performed by an independent investigator blinded to the volume flow analysis outcomes. Follow up DUS imaging including volume-flow assessment will be set at 24h, 6, and 12 months, while fistulograms with QVA analysis will be performed at 6 and 12 months.
Masking Description: QVA analysis will be performed by an investigator blinded to the volume flow analysis outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volume flow group (Experimental): Consecutive patients undergoing sequential volume flow measurements using percutaneous DUS
  Interventions: Diagnostic Test: Volume flow guided angioplasty

INTERVENTIONS:
Diagnostic Test: Volume flow guided angioplasty — Volume flow measurements using DUS will be obtained at the end of each balloon dilation, at 24 hours, 6 months, and one year after index procedure.

SUMMARY:
This is a pilot study investigating a new concept of intra-procedural percutaneous duplex ultrasound (DUS) volume flow-guided balloon angioplasty for the quantification and optimization of endovascular treatment outcomes of dysfunctional autologous arteriovenous fistulae (AVF).

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm clinical trial introducing a new functional index of clinical success of endovascular treatment and investigating the feasibility of volume flow-guided balloon angioplasty of dysfunctional AVF assessed with intraprocedural percutaneous DUS. The study will include consecutive patients undergoing fluoroscopically-guided percutaneous balloon angioplasty due to dysfunctional AVF in the investigator's center. Exclusion criteria will be: (i) not available volume flow values at the time of AVF maturation, (ii) patients with arteriovenous synthetic grafts. Patients' demographical data, dialysis access history, and procedural details will be recorded. Intraprocedural volume flow measurements will be obtained just prior to the procedure and after each balloon dilation. Volume flow measurements will be correlated with digital subtraction angiography quantitative vessel analysis (QVA) performed by an independent investigator blinded to the volume flow analysis outcomes. Follow up DUS imaging including volume-flow assessment will be set at 24h, 6, and 12 months after the index procedure, while fistulograms with QVA analysis will be performed at 6 and 12 months. All DUS measurements will be performed using the same imaging protocol and the same operator. The study's primary endpoints will be (i) the quantification of angioplasty outcome using sequential DUS volume flow analysis following each balloon catheter dilation and (ii) to assess the correlation between volume flow and clinical success defined as high-quality dialysis for a period of at least one month. Secondary endpoints will be (i) re-intervention-free interval defined as the time interval between endovascular treatment and reintervention due to dysfunction recurrence of the treated AVF and (ii) correlation between volume flow and QVA measurements.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing fluoroscopically-guided percutaneous balloon angioplasty due to dysfunctional AVF
* Signed consent form
* Agree to the imaging protocol

Exclusion Criteria:

* not available volume flow values at the time of AVF maturation
* patients with arteriovenous synthetic grafts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Quantification of angioplasty outcome | At the end of the procedure
  The quantification of angioplasty outcomes will be performed using sequential DUS volume flow analysis
Duplex Ultrasound volume flow values achieved following angioplasty and clinical success | 1 month
  The investigators will use ROC analysis to define a cut off value of volume flow increase (ml per minute) at the end of the procedure to predict clinical success.

SECONDARY OUTCOMES:
Re-intervention-free interval | 6 months
  The time interval between endovascular treatment and reintervention due to dysfunction recurrence of the treated AVF
Comparison of Duplex Ultrasound volume flow values with digital subtraction angiography QVA measurements. | 6 months
  To assess wheather a significant volume flow decrease of >50% measured by Duplex ultrasound indicates an analougously significant late lumen loss (mm) of the target lesion measured with QVA analysis of digital subtracted venography

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Spiliopoulos, MD, PhD, EBIR, Principal Investigator — ATTIKO University Hospital
Locations (3):
- Greece (3):
  - "Attikon" University General Hospital, Athens, Attica
  - Medifil SA Hemodialysis Centre, Athens, Attica
  - Nefrologiki SA Hemodialysis Centre, Athens, Attica

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to make individual participant data (IPD) available to other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the publication of the study, indefinitely
Access Criteria: Other researchers upon request